CLINICAL TRIAL: NCT04678856
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Dupilumab in Patients With Uncontrolled, Chronic Rhinosinusitis Without Nasal Polyposis (CRSsNP)
Brief Title: Dupilumab in CRSsNP
Acronym: Liberty CRSsNP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16723; U1111-1246-7522 (Registry Identifier: ICTRP); 2020-003117-35 (EudraCT Number)
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Chronic Rhinosinusitis Without Nasal Polyps; Sinusitis; Chronic Sinusitis; Sinus Disorder; Respiratory Disorder
MeSH Terms: conditions — Sinusitis; Paranasal Sinus Diseases; Respiration Disorders | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part A and B: Dupilumab (Experimental): Participants received dupilumab 300 milligrams (mg) via SC injection q2w for up to 53.1 weeks.
  Interventions: Drug: Dupilumab SAR231893
- Part A and B: Matching placebo (Placebo Comparator): Participants received matching placebo via SC injection q2w for up to 53.2 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dupilumab SAR231893 — Pharmaceutical form:Injection solution Route of administration: Subcutaneous
  Arms: Part A and B: Dupilumab
Drug: Placebo — Pharmaceutical form:Injection solution Route of administration: Subcutaneous
  Arms: Part A and B: Matching placebo

SUMMARY:
Primary Objective:

To evaluate the efficacy of dupilumab as assessed by the reduction at Week 24 in sinus opacification on computerized tomography (CT) scan in the dupilumab group only

Secondary Objectives:

* To evaluate the efficacy of dupilumab as assessed by the reduction at Week 24 in sinus opacification on CT scan and sinus total symptom score (sTSS) compared to placebo
* To evaluate the safety and tolerability of dupilumab in CRSsNP patients compared to placebo
* To evaluate the pharmacokinetics (PK) of dupilumab in CRSsNP patients compared to placebo
* Assessment of immunogenicity to dupilumab over time compared to placebo

DETAILED DESCRIPTION:
The duration of study for each participant will include 2-4 weeks of screening period, 24-52 weeks randomized investigational medicinal product (IMP) intervention period and 12 weeks of follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age at the time of signing the informed consent form (ICF).
* Participants must have bilateral inflammation of paranasal sinuses in CT scan with LMK ≥8 and bilateral ethmoid opacification before randomization.
* Participants must have ongoing symptoms of loss of smell and rhinorrhea (anterior/posterior) of any severity, with or without facial pain/pressure for at least 12 consecutive weeks by Visit 1.
* Participants must have ongoing symptoms of nasal congestion (NC)/obstruction at least 12 consecutive weeks before Visit 1 and a NC score of ≥ 2 at Visit 1 (day score) and Visit 2 (weekly average score).
* Participants must have sTSS (NC, rhinorrhea, facial pain/pressure) ≥5 at Visit 1 (day score) and Visit 2 (weekly average score).
* Participants must have one of the 2 following features:

  * Prior sinonasal surgery (see note at end of section 5.2 for definitions of sinonasal surgery) for CRS,
  * Treatment with systemic corticosteroids (SCS) therapy for CRS as defined by any dose and duration within the prior 2 years before screening (Visit 1) or intolerance/contraindication to SCS.

Exclusion Criteria:

* Participants with nasal conditions/concomitant nasal diseases such as nasal polyposis in endoscopy at Visit 1 or with history of nasal polyposis etc., making them non-evaluable at Visit 1 or for the primary efficacy
* Nasal cavity malignant tumor and benign tumors.
* Forced expiratory volume (FEV1) ≤50% of predicted normal at Visit 1.
* Radiologic suspicion or confirmed invasive or expansive fungal rhinosinusitis.
* Severe concomitant illness(es) that, in the investigator's judgment, would adversely affect participation in the study
* Active tuberculosis or non-tuberculous mycobacterial infection, or a history of incompletely treated tuberculosis unless documented adequately treated.
* Diagnosed active endoparasitic infections; suspected or high risk of endoparasitic infection
* Known or suspected immunodeficiency
* History of malignancy within 5 years before Visit 1, except completely treated in situ carcinoma of the cervix, and completely treated and resolved nonmetastatic squamous or basal cell carcinoma of the skin.
* Active chronic or acute infection requiring treatment with systemic antibiotics, antivirals, or antifungals within 2 weeks before the Screening Visit 1 or during the screening period.
* History of systemic hypersensitivity or anaphylaxis to dupilumab or any of its excipients.
* Participants in prior dupilumab clinical trial or have been treated with commercially available dupilumab within 12 months or who discontinued dupilumab use due to adverse event.
* Participants who are treated with intranasal corticosteroid drops; intranasal steroid emitting devices/stents; nasal spray using exhalation delivery system, such as Xhance™, during screening period.
* Participants on unstable dose of intranasal corticosteroids (INCS) spray 4 weeks prior to Screening Visit (Visit1) and during screening period.
* Participants who have undergone sinus intranasal surgery (including polypectomy) within 6 months prior to Visit 1.
* Participants who have taken:

  * Biologic therapy/systemic immunosuppressant to treat inflammatory disease or autoimmune disease within 5 half-lives prior to Visit 1
  * Any investigational mAb within 5 half-lives prior to Visit 1
  * Anti-IgE therapy (omalizumab) within 4 months prior to Visit 1.
* Treatment with a live (attenuated) vaccine within 4 weeks prior to Visit 1
* Leukotriene antagonists/modifiers unless participant is on a continuous treatment for at least 30 days prior to Visit 1.
* Initiation of allergen immunotherapy within 3 months prior to Visit 1 or a plan to begin therapy or change its dose during the screening or treatment period.
* Participants received SCS during screening period (between Visit 1 and Visit 2).
* Either intravenous immunoglobulin therapy and/or plasmapheresis within 30 days prior to Screening Visit (Visit 1).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (58):
- United States (11):
  - Sacramento Ear, Nose & Throat Site Number : 8400010, Roseville, California
  - Bensch Clinical Research LLC Site Number : 8400015, Stockton, California
  - Colorado Allergy and Asthma Centers, PC Site Number : 8400003, Denver, Colorado
  - University of Missouri Health System Site Number : 8400016, Columbia, Missouri
  - Nebraska Medical Research Institute Site Number : 8400007, Papillion, Nebraska
  - Optimed Research, LTD Site Number : 8400017, Columbus, Ohio
  - Vital Prospects Clinical Research Institute, P.C. Site Number : 8400004, Tulsa, Oklahoma
  - Essential Medical Research, LLC Site Number : 8400014, Tulsa, Oklahoma
  - Pharmaceutical Research & Consulting, Inc. Site Number : 8400006, Dallas, Texas
  - Alamo ENT Associates Site Number : 8400021, San Antonio, Texas
  - Eastern Virginia Medical School (EVMS) Medical Group - Otola Site Number : 8400009, Norfolk, Virginia
- Argentina (3):
  - Investigational Site Number : 0320002, Buenos Aires
  - Investigational Site Number : 0320003, Ciudad Autonoma Buenos Aires
  - Investigational Site Number : 0320001, Ciudad Autonoma Buenos Aires
- Belgium (2):
  - Investigational Site Number : 0560002, Ghent
  - Investigational Site Number : 0560001, Leuven
- Canada (9):
  - Investigational Site Number : 1240013, Vancouver, British Columbia
  - Investigational Site Number : 1240010, Hamilton, Ontario
  - Investigational Site Number : 1240007, Kingston, Ontario
  - Investigational Site Number : 1240016, London, Ontario
  - Investigational Site Number : 1240001, Montreal, Quebec
  - Investigational Site Number : 1240012, Montreal, Quebec
  - Investigational Site Number : 1240002, Trois-Rivières, Quebec
  - Investigational Site Number : 1240005, Québec
  - Investigational Site Number : 1240003, Québec
- Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago, Chile
- China (6):
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560005, Changchun
  - Investigational Site Number : 1560013, Changsha
  - Investigational Site Number : 1560010, Chongqing
  - Investigational Site Number : 1560006, Shanghai
  - Investigational Site Number : 1560008, Yantai
- Hungary (2):
  - Investigational Site Number : 3480004, Budapest
  - Investigational Site Number : 3480001, Pécs
- Portugal (3):
  - Investigational Site Number : 6200002, Aveiro
  - Investigational Site Number : 6200001, Guimarães
  - Investigational Site Number : 6200003, Matosinhos Municipality
- Russia (4):
  - Investigational Site Number : 6430005, Moscow
  - Investigational Site Number : 6430002, Saint Petersburg
  - Investigational Site Number : 6430003, Saint Petersburg
  - Investigational Site Number : 6430001, Stavropol
- South Korea (2):
  - Investigational Site Number : 4100003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 4100002, Seoul, Seoul-teukbyeolsi
- Spain (8):
  - Investigational Site Number : 7240002, Seville, Andalusia
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240007, Santander, Cantabria
  - Investigational Site Number : 7240004, Jerez de la Frontera, Cádiz
  - Investigational Site Number : 7240009, Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240005, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240008, Pamplona, Navarre
  - Investigational Site Number : 7240010, Madrid
- Investigational Site Number : 7520001, Stockholm, Sweden
- Ukraine (6):
  - Investigational Site Number : 8040005, Dnipro
  - Investigational Site Number : 8040001, Ivano-Frankivsk
  - Investigational Site Number : 8040004, Kharkiv
  - Investigational Site Number : 8040008, Kyiv
  - Investigational Site Number : 8040002, Kyiv
  - Investigational Site Number : 8040007, Kyiv

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16723 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25252&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 57 centers in 13 countries. A total of 269 participants were screened between 02 December 2020 to 26 April 2023, of which 198 participants were screen failures. Screen failures were mainly due to not meeting the eligibility criteria.
Pre-assignment Details: A total of 71 participants were randomized in a ratio of 1:1 to receive dupilumab or matching placebo. Randomization was stratified by screening blood eosinophil count (≥300 cells per cubic millimeter [/mm^3] or <300 cells/mm^3), background intranasal corticosteroids (INCS) use (yes or no), and region.
Groups:
- Placebo: Participants received matching placebo via subcutaneous (SC) injection every 2 weeks (q2w) for up to 53.2 weeks.
- Dupilumab 300 mg q2w: Participants received dupilumab 300 milligrams (mg) via SC injection q2w for up to 53.1 weeks.
Period: Overall Study
Arm/Group | Placebo | Dupilumab 300 mg q2w
Started | 33 | 38
Completed | 25 | 37
Not Completed | 8 | 1
Not completed — Not related to Coronavirus Disease-2019 (COVID-19) | 3 | 0
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants with a treatment kit number allocated and recorded in the interactive response technology (IRT) database, and regardless of whether the treatment kit was used or not.
Groups:
- Placebo: Participants received matching placebo via SC injection q2w for up to 53.2 weeks.
- Dupilumab 300 mg q2w: Participants received dupilumab 300 mg via SC injection q2w for up to 53.1 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | Dupilumab 300 mg q2w | Total
Number analyzed (Participants) | 33 | 38 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.45 (17.46) | 46.45 (12.60) | 46.92 (14.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 25 | 41
  Male | 17 | 13 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 30 | 31 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Lund-Mackay (LMK) Score [Mean (Standard Deviation); unit: Score on a scale] | 11.50 (3.19) | 11.41 (3.69) | 11.45 (3.44)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Opacification of Sinuses Assessed by Computed Tomography (CT) Scan Using the Lund Mackay (LMK) Score in Dupilumab Group
Description: The CT scan LMK staging system represented the most widely established method of sinus CT scoring. The LMK total score is based on assessment of the CT scan findings for each sinus area (maxillary, anterior ethmoid, posterior ethmoid, sphenoid, and frontal sinus on each side). The extent of mucosal opacification is rated on a 3-point scale ranging from 0 = normal to 2 = total opacification. In addition, the ostiomeatal complex is graded as 0 = not occluded or 2 = occluded. The maximum score is therefore 12 per side; total score ranges from 0 (normal) to 24 (more opacified), corresponding to the sum of all sinuses and the ostiomeatal unit. Higher score indicated worse outcome. Baseline was defined as the last available value up to randomization date and prior to the first dose of study medication.
Time Frame: Baseline (Day 1) and Week 24
Population: Intent-to-treat (ITT) population with screening blood eosinophil count ≥300 cells/mm^3 included all randomized participants with screening blood eosinophil count ≥300 cells/mm^3 analyzed according to the treatment group allocated by randomization regardless if treatment kit was used or not.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Dupilumab 300 mg q2w
Number analyzed (Participants) | 16
Score on a scale | -6.63 (3.91)

2. Secondary Outcome: Change From Baseline to Week 24 in Opacification of Sinuses Assessed by CT Scan Using the LMK Score
Description: as for outcome 1
Time Frame: Baseline (Day 1) and Week 24
Population: ITT population with screening blood eosinophil count ≥300 cells/mm^3 included all randomized participants with screening blood eosinophil count ≥300 cells/mm^3 analyzed according to the treatment group allocated by randomization regardless if treatment kit was used or not. Only those participants with data collected at Week 24 are reported.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 14 | 16
Score on a scale | -0.68 (2.26) | -6.63 (3.91)

3. Secondary Outcome: Change From Baseline to Week 24 in Sinus Total Symptom Score (sTSS)
Description: The sTSS is a composite score derived from the following individual items: nasal congestion (NC), anterior/posterior rhinorrhea, and facial pain/pressure. Each of the individual items were scored from 0 (no symptoms) to 3 (severe symptoms). The total score ranges from 0 to 9 and consists of the sum of NC, the averaged rhinorrhea item scores, and facial pain/pressure scores. Higher scores on sTSS indicated greater overall symptom severity. Baseline was defined as the last available value up to randomization date and prior to the first dose of study medication.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 14 | 16
Score on a scale | -1.75 (2.19) | -3.18 (2.68)

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious AEs (TESAEs), and TEAEs Leading to Treatment Discontinuation
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were AEs that developed, worsened or became serious during the treatment-emergent period. A SAE was defined as any untoward medical occurrence that, at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: From the first dose of study drug (Day 1) up to the last dose of study drug administration (373 days) + 98 days, up to 471 days
Population: Safety population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 33 | 38
Participants
  TEAEs | 27 | 29
  TESAEs | 6 | 3
  TEAEs leading to treatment discontinuation | 0 | 1

5. Secondary Outcome: Serum Concentration of Dupilumab Over Time
Description: Blood samples were collected at the specified timepoints to evaluate serum concentration of dupilumab.
Time Frame: Baseline (Day 1) and Weeks 12, 24 and 52
Population: Pharmacokinetic (PK) population included all participants in the safety population with at least 1 non-missing result for functional dupilumab concentration in serum after the first dose of the study intervention. Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | Dupilumab 300 mg q2w
Number analyzed (Participants) | 28
Nanograms per milliliter
  Baseline: number analyzed (Participants) | 22
  Baseline | 0.00 (0.00)
  Week 12: number analyzed (Participants) | 25
  Week 12 | 54733.20 (26222.53)
  Week 24 | 62192.86 (23979.23)
  Week 52: number analyzed (Participants) | 20
  Week 52 | 68365.00 (30613.86)

6. Secondary Outcome: Number of Participants With Antidrug Antibody (ADA) Response to Dupilumab and Positive Neutralizing Antibody (Nab)
Description: Plasma samples were collected to evaluate antibodies to dupilumab. Pre-existing immunoreactivity was defined as an ADA positive response in the assay at baseline with all post first dose ADA results negative, OR an ADA positive response at baseline with all post first dose ADA responses less than 4-fold over baseline titer levels. Treatment-emergent ADA responses were defined as a positive response in the ADA assay post first dose, when baseline results were negative or missing. Treatment-boosted response was defined as an ADA positive response in the assay post first dose that was greater-than or equal to 4-fold over baseline titer levels, when baseline results were positive. Samples positive in the ADA assay were further characterized for the presence of NAbs.
Time Frame: Baseline (Day 1) and up to Week 52
Population: ADA population included all participants in the safety population who had at least 1 non-missing result in the ADA assay after the first dose of the study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Dupilumab 300 mg q2w
Number analyzed (Participants) | 33 | 38
Participants
  Pre-existing immunoreactivity | 1 | 0
  Treatment-emergent ADA response | 1 | 1
  Treatment-boosted ADA response | 1 | 0
  Positive Nab | 3 | 1

ADVERSE EVENTS:
Time Frame: TEAEs and TESAEs were collected from the first dose of study drug (Day 1) up to the last dose of study drug administration (373 days) + 98 days, up to 471 days. All-cause mortality (deaths) were collected from participant's screening (Day -28) to the end of follow-up for each participant, up to 476 days.
Description: Analysis was performed on safety population.
Arm/Group | Placebo | Dupilumab 300 mg q2w
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/38
Serious Adverse Events (participants affected / at risk) | 6/33 | 3/38
Other Adverse Events (participants affected / at risk) | 12/33 | 20/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | Dupilumab 300 mg q2w (N=38)
Myocardial Bridging (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Chronic Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Biloma (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diabetic Neuropathy (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | Dupilumab 300 mg q2w (N=38)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (3)
Injection Site Erythema (General disorders) | 1 (20) | 4 (9)
Injection Site Reaction (General disorders) | 1 (8) | 3 (12)
Injection Site Swelling (General disorders) | 2 (23) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Covid-19 (Infections and infestations) | 7 (8) | 8 (9)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (3)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (3)
Otitis Media (Infections and infestations) | 1 (1) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 2 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT04678856/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT04678856/SAP_001.pdf